CLINICAL TRIAL: NCT04075240
Title: Extended Venous Thromboembolism Prophylaxis Comparing Rivaroxaban and Aspirin to Aspirin Alone Following Total Hip and Knee Arthroplasty (EPCATIII)
Brief Title: VTE Prevention Following Total Hip and Knee Arthroplasty
Acronym: EPCATIII
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sudeep Shivakumar (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Nova Scotia Health Authority (Other); Canadian Venous Thromboembolism Clinical Trials and Outcomes Research (CanVECTOR) Network (Network)
Responsible Party: Sponsor-Investigator, Sudeep Shivakumar, Head, Division of Hematology, Nova Scotia Health Authority
Organization: Nova Scotia Health Authority (Other)
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: EPCATIII.001
Record Dates: First submitted 2019-08-29; First posted 2019-08-30 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Venous Thromboembolism
Keywords: total hip and knee arthroplasty
MeSH Terms: conditions — Venous Thromboembolism | interventions — Rivaroxaban; Aspirin

STUDY DESIGN:
Intervention Model Description: randomized, controlled, double-blind
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: over-encapsulated rivaroxaban/ASA
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- THA-control arm (Active Comparator): Total Hip Arthroplasty: 5 days of rivaroxaban, followed by 30 days of aspirin
  Interventions: Drug: Rivaroxaban 10 MG and acetylsalicylic acid 81 mg
- THA-study arm (Experimental): Total Hip Arthroplasty: 35 days of aspirin
  Interventions: Drug: acetylsalicylic acid 81 mg
- TKA-control arm (Active Comparator): Total Knee Arthroplasty: 5 days of rivaroxaban, followed by 9 days of aspirin
  Interventions: Drug: Rivaroxaban 10 MG and acetylsalicylic acid 81 mg
- TKA-study arm (Experimental): Total Knee Arthroplasty: 14 days of aspirin
  Interventions: Drug: acetylsalicylic acid 81 mg

INTERVENTIONS:
Drug: Rivaroxaban 10 MG and acetylsalicylic acid 81 mg — Starting post op, rivaroxaban (5 days) followed by aspirin (9 days for TKA; 30 days for THA)
  Other Names: Xarelto 10mg and aspirin 81mg
  Arms: THA-control arm; TKA-control arm
Drug: acetylsalicylic acid 81 mg — Starting post op, aspirin for 9 days for TKA and 30 days for THA
  Other Names: aspirin 81mg
  Arms: THA-study arm; TKA-study arm

SUMMARY:
Consented patients undergoing elective total hip and total knee arthroplasty will be randomized to receive either aspirin alone or aspirin and rivaroxaban for prevention of venous thromboembolism.

DETAILED DESCRIPTION:
Aspirin and rivaroxaban prevent venous thromboembolism (VTE) via different mechanisms. Aspirin is significantly cheaper than rivaroxaban. Aspirin in combination with rivaroxaban was shown to be safe and efficacious in a non-inferiority trial (EPCATII) when compared to rivaroxaban alone.

This study will assess if aspirin alone is non-inferior to rivaroxaban and aspirin in the prevention of venous thromboembolism.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing elective THA/TKA at the participating institutions will be potentially eligible for this study
2. Written informed consent in accordance with federal, local and institutional guidelines

Exclusion Criteria:

1. Previous documented VTE (proximal DVT or any PE)
2. Hip or lower limb fracture in the previous three months, not related to present surgery
3. Metastatic cancer
4. Life expectancy less than 6 months
5. History of major bleeding that in the judgment of the investigator precludes use of anticoagulant prophylaxis
6. History of aspirin allergy, active peptic ulcer disease or gastritis that in the judgment of investigator precludes use of aspirin
7. History of significant hepatic disease or any other condition that in the judgment of the investigator precludes the use of rivaroxaban
8. Creatinine clearance less than 15 ml per minute
9. Pre-operative platelet count less than 100 x 109 /L
10. Need for long-term anticoagulation due to a pre-existing co-morbid condition or due to the development of VTE following surgery but prior to randomization
11. Received anticoagulation post operatively
12. Bilateral THA/TKA or simultaneous hip and knee arthroplasty
13. Major surgical procedure within the previous 3 months
14. Requirement for major surgery post arthroplasty within a 90 day period
15. Chronic daily aspirin use with dose greater than 100 mg a day
16. Women of childbearing potential who are not abstinent or do not use effective contraception or are breast-feeding throughout the study drug period
17. Unwilling or unable to give consent
18. Previous participation in the EPCAT III study
19. Under 18 years of age
20. Concomitant use of drugs that are strong inhibitors of P-gp AND CYP3A4 (e.g., systemic treatment with ketoconazole, itraconazole, or ritonavir) or strong inducers of P-gp AND CYP3A4 (e.g., rifampicin, phenytoin, carbamazepine, phenobarbital, St. John's Wort)
21. Known allergy to food dye

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5400 (Estimated)
Dates: Start 2021-02-04 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Venous thromboembolism | 90 days
  symptomatic proximal deep vein thrombosis or pulmonary embolism
Bleeding | 90 days
  major and clinically relevant, non-major bleeds

SECONDARY OUTCOMES:
Survival | 90 days
  all cause death
Cost-effectiveness | 90 days
  quantitatively describe the costs of symptomatic thromboembolism events and major bleeding episodes

CONTACTS AND LOCATIONS:
Overall Officials: Sudeep P Shivakumar, MD, Principal Investigator — Dalhousie University/Nova Scotia Health Authority
Locations (1):
- Queen Elizabeth II HSC, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No